CLINICAL TRIAL: NCT01141205
Title: Phase I Study: HIV-1 Peptide Immunisation of Individuals in West Africa to Prevent Disease
Brief Title: HIV-1 Peptide Immunisation of Individuals in West Africa to Prevent Disease
Acronym: HIV-BIS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Statens Serum Institut (Other)
Collaborators: Ministry of the Interior and Health, Denmark (Other Government); European and Developing Countries Clinical Trials Partnership (EDCTP) (Other Government)
Responsible Party: Principal Investigator, Anders Fomsgaard, Chief Medical Doctor, Statens Serum Institut
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HIV-BIS NCP03/2009; EDCTP_MSI.2009.10800.001 (Other Grant/Funding Number: EDCTP_MSI.2009.10800.001)
Record Dates: First submitted 2010-06-09; First posted 2010-06-10 (Estimated); Results first posted 2012-10-15 (Estimated); Last update posted 2013-08-08 (Estimated); Status verified 2013-08

CONDITIONS: Aids, Cdc Group I
Keywords: AIDS vaccines; HIV-1 vaccine; Therapeutic vaccine; Cellular immunity
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- AFO-18 (Experimental): 18 peptides representing CD8 and CD4 epitopes mainly on HIV-1 in an adjuvants (CAF01)
  Interventions: Biological: AFO-18
- Saline (Placebo Comparator): Saline
  Interventions: Drug: Saline

INTERVENTIONS:
Biological: AFO-18 — 18 peptides representing CD8 and CD4 epitopes mainly on HIV-1 in an adjuvants (CAF01)
  Other Names: CAF01; HIV-1 peptides
  Arms: AFO-18
Drug: Saline — 1.2 ml saline intramuscularly
  Other Names: NaCl
  Arms: Saline

SUMMARY:
Treatment: Immunization with peptide-mix and adjuvant. The vaccine should induce cellular immunity against HIV-1.

Target group: Untreated healthy individuals with chronic HIV-1 infection.

Purpose: The primary purpose is to evaluate tolerability and safety of the vaccine.

The secondary purpose is to evaluate the clinical effect of the vaccination treatment as measured by induction of immunity, lowering of viral load, induction of escape mutations in the virus and improvement in the patient CD4 lymphocyte blood counts.

The third purpose is to evaluate the feasibility of conducting a therapeutic HIV immunization study in a poorly-resourced African setting.

Design: The experiment is designed as a blinded, placebo-controlled phase 1 clinical trial in HIV-1 infected individuals in West Africa.

Numbers of individuals: Phase I: 20 fully evaluable HIV-1-infected patients should enter the study (15 vaccine treated and 5 placebo(saline) treated controls).

DETAILED DESCRIPTION:
The HIV infection does not leave lifelong immunity, but leads to break down of the immune system, opportunistic infections and death. The immunity obtained by the infection itself can only partially contain the HIV infection. The purpose with a targeted therapeutic vaccination is therefore in addition to the existing immunity to induce a broader, more powerful and more rationally or better directed immunity than the one induced by the "natural" HIV-1 infection. This would potentially lower the viral load in the blood making it more difficult to spread the virus to others and prolong the time to AIDS disease and medical treatment. There is a need for new rational vaccination possibilities, able to prevent (HIV) disease, postpone the need for antiretroviral medical treatment, prolong the life, and limit spread of HIV-1 in the population. The present protocol seak to introduce such a new immune treatment principle for HIV-1 infected individuals. In this study, individuals with chronic HIV-1 infection will be vaccinated with selected synthetic HIV immune-peptides representing new discovered conserved target´s on the virus. The vaccine should induce new immunity against several epitope targets on their HIV, whereby the HIV infection may be controlled for a longer time by the immune system. The purpose of the study is primarily to evaluate the safety and tolerability of the vaccine and secondary to evaluate the immunological and antiviral response in the vaccinated individuals.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 seropositive with measurable viral load >10e3 copies/ml and CD4+ T-cell count >400 CD4+ cells/µl.
2. Not in Antiretroviral Therapy (>1 year).
3. Male or female with age between 18 and 50 years.
4. Normal values for the area of liver and kidney enzymes, blood cell count with differential counts (e.g. white blood cells, lymphocytes, platelets/thrombocytes) and Hemoglobin
5. Expected to follow the instructions.
6. Written informed consent after oral and written information.

Exclusion Criteria:

1. Vaccinated with other vaccines within 3 months before the first vaccination.
2. Treated with immune modulating medicine within 3 month before the first immunization.
3. Other important active chronic infectious diseases likely to influence the HIV-1 infection, like HIV-2, HBV, HCV and TB
4. Significant medical disease as judged by the investigators, for example severe asthma/COLD, badly regulated heart disease, insulin-dependent diabetes mellitus.
5. Severe allergy or earlier anaphylactic reactions.
6. Active autoimmune diseases.
7. Simultaneous treatment with other experimental drugs.
8. Laboratory parameters outside the 'normal' range for the area and which are considered clinically significant.
9. Pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2009-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anders Fomsgaard, DMSc, Study Director — Statens Serum Institut; Zacarias Jose da Silva, PhD, Principal Investigator — Bandim Health Project, Bissau, Guinea-Bissau
Locations (2):
- Guinea-Bissau (2):
  - Hospital Nacional Simao Mendes, Bissau, Guinea-Bissau
  - Hospital Nacional Simao Mendes, Bissau

REFERENCES:
- [Result] Roman VR, Jensen KJ, Jensen SS, Leo-Hansen C, Jespersen S, da Silva Te D, Rodrigues CM, Janitzek CM, Vinner L, Katzenstein TL, Andersen P, Kromann I, Andreasen LV, Karlsson I, Fomsgaard A. Therapeutic vaccination using cationic liposome-adjuvanted HIV type 1 peptides representing HLA-supertype-restricted subdominant T cell epitopes: safety, immunogenicity, and feasibility in Guinea-Bissau. AIDS Res Hum Retroviruses. 2013 Nov;29(11):1504-12. doi: 10.1089/AID.2013.0076. Epub 2013 Jun 21. PMID 23634822

RESULTS

PARTICIPANT FLOW:
Recruitment Details: medical clinic
Groups:
- AFO-18: 18 peptides representing 15 CD8 and 3 CD4 epitopes on HIV-1 plus 1 CD4 T helper epitope unrelated to HIV in an adjuvant (CAF01). Total 4.5 mg peptide (250 micro gram of each peptide) in CAF01 adjuvant. Total volume of 1.25 ml was injected i.m. (in m. deltoideus) at weeks 0, 2, 4, 8
- Saline: Placebo was Sterile saline injection, 1.25 ml i.m. (in m. deltoideus) at each vaccination weeks 0, 2, 4, 8
Period: Overall Study
Arm/Group | AFO-18 | Saline
Started | 18 | 5
Completed | 15 | 3
Not Completed | 3 | 2
Not completed — Physician Decision | 1 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Saline: Saline injection
- Total: Total of all reporting groups
Arm/Group | AFO-18 | Saline | Total
Number analyzed (Participants) | 18 | 5 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 5 | 23
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 34 (2) | 29 (2) | 32 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 3 | 20
  Male | 1 | 2 | 3
Region of Enrollment [Number; unit: participants]
  Guinea-Bissau | 18 | 5 | 23

OUTCOME MEASURES:

1. Primary Outcome: Tolerability and Safety of the Treatment.
Description: We report here the numbers of participants with vaccine related adverse events degree 3 or 4.
  Our goal for safety and tolerability was: "Fewer than or 3 patients of the 15 vaccine treated show treatment related (reaction 3) side-effects of degree 3 or 4".
Time Frame: up to 6 months after end of treatment
Population: Analyzed: number of participants started minus individuals lost to follow up or participants that withdraw. Thus we include the two individuals where the physician stopped his/her participation because of SAE not related to the vaccine or to the placebo. Reported: numbers of participants with vaccina related SAE
Measure: Number; unit: participants
Groups:
- Vaccinee: participants receiving active peptide in CAF01 adjuvants vaccine
- Placebo: participants receiving saline
Arm/Group | Vaccinee | Placebo
Number analyzed (Participants) | 16 | 4
participants | 0 | 0

2. Secondary Outcome: Induction of New T-cell Immune Response by the Vaccine
Description: induction of new T-cell immune response against one or more of the vaccine epitopes using Interferon gamma Enzyme Linked Immuno spot assay (IFNg-ELISPOT assay)measuring Spot forming Unis per 1 million periferal blood mononuclear cells (SFU/1 mio PBMCs) above treshold (> 50 sfu/mio PBMC).
Time Frame: up to 6 months after last immunisation
Population: Analyzed: Participants minus drop-outs and withdrawn participants. Reported: numbers of participants with a new induced ELISPOT Y-cell immune response to the vaccine peptide epitopes
Measure: Number; unit: ELISPOT responders
Groups:
- Placebo Saline: Saline injection
Arm/Group | AFO-18 | Placebo Saline
Number analyzed (Participants) | 14 | 2
ELISPOT responders | 6 | 0

3. Secondary Outcome: Lowering of HIV-1 RNA Viral-load in HIV-1 Immune Responders More Than 1 Log
Description: changes (lowering) in Plasma HIV-1 RNA viral-load (measured by Quantitative RT-PCR kit, ROCHE) of more than 1 log
Time Frame: up to 6 months post immunization
Population: Participants minus drop outs and participants withdrawn by them selves or by the physicians
Measure: Number; unit: participants with lowering of VL
Groups:
- Vaccinee: participants receiving active HIV-1 peptide vaccine in CAF01 adjuvant i.m.
- Saline: Placebo participants receiving sterile saline i.m.
Arm/Group | Vaccinee | Saline
Number analyzed (Participants) | 15 | 3
participants with lowering of VL | 0 | 0

4. Secondary Outcome: Increase in Blood CD4 T-cell Counts
Description: Analyzed: Participants (minus drop-outs and withdrawn) with measured blood CD4 T-cell counts (cells/microliter). Reported: Numbers of participants obtaining an increase in measured blood CD4 T-cell counts post vaccination of >100 CD4 Tcell per microliter
Time Frame: up to 6 months post vaccination
Population: Participants minus drop-outs and withdrawn participants
Measure: Number; unit: participants with increased CD4 count
Arm/Group | Vaccinee | Placebo
Number analyzed (Participants) | 15 | 3
participants with increased CD4 count | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: One participant in the vaccinee group of 18 individuals had a SAE (serious infection) not related to the vaccine. One participant in the saline placebo group of 5 individuals experienced a SAE (increase in liver enzymes) not related to the placebo saline.
  None others experienced any AE was noted.
Arm/Group | AFO-18 | Saline
Serious Adverse Events (participants affected / at risk) | 1/18 | 1/5
Other Adverse Events (participants affected / at risk) | 0/18 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AFO-18 (N=18) | Saline (N=5)
Died of pneumonia (Infections and infestations) | 1 (1) | 0 (0) — One participant died of severe gastroenteritis and pneumonia unrelated to the vaccine
Increase in liver enzymes (Infections and infestations) | 0 (0) | 1 (1) — One placebo (saline) participant got elevation of liverenzymes (unrelated to the placebo)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes